CLINICAL TRIAL: NCT01763697
Title: Taste Acuity and Caloric Intake After Acute Morphine Administration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Denis Antoine, Instructor, Johns Hopkins University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: NA_00046407; K24DA023186-06 (NIH)
Record Dates: First submitted 2013-01-07; First posted 2013-01-09 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Taste Sweet; Taste Salty; Feeding Behavior
Keywords: Taste acuity; Feeding behavior; opioid; Quantitative assessment
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Morhpine/Taste acuity (Active Comparator): Taste acuity assessment after 1mg subcutaneous morphine injection
  Interventions: Behavioral: taste acuity assessment; Behavioral: Recorded meal
- Placebo/Taste acuity (Placebo Comparator): Taste acuity assessment after subcutaneous placebo injection
  Interventions: Behavioral: taste acuity assessment; Behavioral: Recorded meal
- Morphine4/Taste acuity (Active Comparator): Taste acuity assessment after 4mg subcutaneous morphine injection
  Interventions: Behavioral: taste acuity assessment; Behavioral: Recorded meal

INTERVENTIONS:
Behavioral: taste acuity assessment — Quantitative measurement of for tasting detection and recognition thresholds, magnitude of perception and hedonic response.
Behavioral: Recorded meal

SUMMARY:
This study will investigate the effects of acute morphine administration on taste acuity and how much a person eats. It is hypothesized that there will be a dose dependent decrease in taste acuity and dose dependent increase in food intake associated with acute morphine administration. Knowledge from this study will impact the future of feeding behavior and obesity research in the general population. Results will also promote exploration of the long-term effect of opioid abuse on taste acuity and feeding behavior in substance abusing populations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male and female volunteers
* Ages of 18 to 65

Exclusion Criteria:

* History of drug dependence (including opioid use disorders)
* History of taste dysfunction
* Significant medical or Axis I psychiatric disorder
* Any trauma or surgical procedures to the head or neck region
* Medication or illicit drug more than 4 out of the last 30 days.
* Pregnancy
* Abnormal electrocardiogram findings
* Negative rating of greater than 40% of the foods available for consumption

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Taste | 3 hours after dose administration
  The primary outcome variable will be the taste acuity profile, which includes the taste detection threshold, recognition threshold, magnitude estimation, and hedonic response.

SECONDARY OUTCOMES:
Calories | 6 hours after dose administration
  The secondary outcome measure will be the amount of calories consumed over a 2 hours period following the drug administration.

CONTACTS AND LOCATIONS:
Overall Officials: Denis G Antoine, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States